CLINICAL TRIAL: NCT05781451
Title: A Phase 2, Open Label Study of Anti-BTLA Agonist Therapy in Subjects With Primary Sjogren's Syndrome
Brief Title: Anti-BTLA Agonist Therapy in Subjects With Primary Sjogren's Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug unavailable
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Matthew C. Baker, Clinical Chief and Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68283
Record Dates: First submitted 2023-02-23; First posted 2023-03-23 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Primary Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3361237 (Experimental): All patients will receive LY3361237 450mg subcutaneously every 2 weeks for a total of 12 weeks.
  Interventions: Drug: LY3361237

INTERVENTIONS:
Drug: LY3361237 — All patients will receive LY3361237 450mg subcutaneously every 2 weeks for a total of 12 weeks.
  Other Names: Venanprubart

SUMMARY:
This will be a single-site, open-label study in patients with primary Sjogren's syndrome. The aim of this clinical trial is to evaluate the safety and efficacy of anti-BTLA agonist therapy (LY3361237) in treating patients with primary Sjogren's syndrome.

The primary objective is to evaluate the efficacy of LY3361237 in patients with primary Sjogren's syndrome by assessing changes in the Sjogren's Tool for Assessing Response (STAR) after 12 weeks of treatment.

The secondary objective is to determine the effect of LY3361237 on glandular changes measured by PET/MRI.

DETAILED DESCRIPTION:
This study is a single-site, open-label study in subjects with primary Sjogren's syndrome being conducted at the Stanford University rheumatology clinic. All eligible subjects will receive LY3361237 450mg SC Q2W over a period of 12 weeks and will be followed up for an additional 10 weeks after the last dose. Twelve subjects will be included in the study.

After the Screening visit, consenting patients will be seen in clinic on day 1 (Baseline) and return to clinic on Weeks 2, 4, 6, 8, 10, 12, and 22.

At Screening (up to 35 days before baseline), a complete medical history, physical exam, vital signs, clinical laboratory tests [comprehensive metabolic panel, complete blood count, quantitative immunoglobulins, ANA, RF, anti-Ro, anti-La, C3, C4, ESR, CRP, urinalysis, urine protein:creatinine, serum pregnancy test for females, HIV serologies, hepatitis B serologies, hepatitis C serologies, quantiFERON test for tuberculosis, SARS-CoV-2 PCR], chest x-ray, electrocardiogram, and salivary gland ultrasound will be conducted.

At all subsequent visits, at a minimum, a complete physical exam, vital signs, focused history, and clinical laboratory tests (comprehensive metabolic panel, complete blood count, ESR, CRP, and urine pregnancy test for females) will be conducted.

Efficacy will be assessed using the Sjogren's Tool for Assessing Response (STAR) and by measuring changes in unstimulated salivary flow rate, changes in salivary glands by ultrasound, changes in salivary glands by PET/MRI, changes in Schirmer I testing, changes in laboratory values including inflammatory markers (ESR, CRP) complement levels (C3, C4), immunoglobulins (IgG, IgA, IgM), and autoantibodies (ANA, SS-A, SS-B, RF), and changes in patient reported outcomes.

At Screening, Baseline, Week 4, and Week 12, patients will record their global assessment of disease as well as visual analog scales for ocular and salivary symptoms and the ESSPRI. At Baseline, Week 4, and Week 12, patients will record the FACIT-F for fatigue and RAND SF-36, and the physician will calculate the ESSDAI, ClinESSDAI, physician global assessment of disease, and tender and swollen joint count.

In addition, safety will be assessed for all patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for enrollment in the study only if they meet all of the following criteria:

* Have given written informed consent
* Are men or women aged 18 to 85, inclusive, at the time of initial screening
* Have a confirmed diagnosis of primary Sjogren's syndrome by the 2016 ACR-EULAR classification criteria for primary Sjogren's syndrome [2]
* ≥50mm on a visual analog scale (VAS) for ocular dryness or oral dryness or ≥5 on the ESSPRI score for dryness
* Have a Hočevar salivary gland ultrasound score (SGUS) (on a 0-48 point scale) and ≥10 [to detect relatively early disease with less anatomic derangement that will potentially be more responsive to treatment and to exclude patients with no changes on ultrasound that would preclude an ability to see improvement] [3]
* All women (regardless of childbearing potential) must test negative for pregnancy at the time of screening. Women must also agree to use a reliable method of birth control from screening until 12 weeks following last dose of study drug (adequate contraceptive measures include: intrauterine devices, hormonal contraceptives, complete sexual abstinence, or vasectomized partner), unless they are not of child-bearing potential as defined by meeting either of the following:

  * Are at least 6 weeks after bilateral oophorectomy, tubal ligation, or hysterectomy
  * Are postmenopausal, as defined by having had spontaneous amenorrhea for at least 12 months and a follicle-stimulating hormone level >40 mIU/mL at screening
* Have venous access sufficient to allow for blood sampling, as per the protocol
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Prior treatment with a BTLA agonist within 6 months before baseline
* Use of other biologic agents including TNF inhibitors, abatacept, IL-6 inhibitors, or BAFF inhibitors within 8 weeks prior to baseline
* Use of a B cell depleting therapy (such as rituximab) within 12 months prior to baseline
* A history of, or current, inflammatory or autoimmune disease (that could affect the interpretation of safety or efficacy outcomes) other than primary Sjogren's syndrome
* Evidence of active tuberculosis, HIV, or hepatitis B or C infection
* Have a diagnosis or history of malignant disease within 5 years prior to baseline, with the following exceptions: basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years and/or cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to baseline
* Prior LASIK or radial keratotomy surgery which could affect symptomatic complaints of eye dryness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Sjogren's Tool for Assessing Response (STAR) | Baseline and Week 12
  Change from Baseline to Week 12 after treatment with LY3361237. STAR is intended to assess treatment efficacy based on improvement of disease activity for primary Sjögren's syndrome. The STAR contains 5 domains: systemic activity, symptoms, lacrimal and glandular gland function, and biomarkers of auto-immune activity.
  The score consists of five domains (systemic activity worth 3 points, patient-reported outcome worth 3 points, lacrimal gland function worth 1 point, salivary gland function worth 1 point, and biological worth 1 point).
  A patient is considered a STAR responder if they accrue ≥5 points.

SECONDARY OUTCOMES:
Change in unstimulated salivary flow | Baseline and Week 12
  Unstimulated salivary flow as assessed by sialometry.
Change in salivary gland ultrasound score | Baseline and Week 12
  The Hočevar salivary gland ultrasound score (SGUS) will be calculated by assessing Parenchymal echogeneity, Homogeneity, Presence of hypoechogenic areas, Hyperechogenic reflections, and Clearness of salivary gland borders. The Hočevar ultrasound score will be calculated by summation of the grades for the five parameters described above for all four glands, with a range of 0-48 (with a higher score reflecting worse disease activity).
Change in MRI findings on PET/MRI imaging | Baseline and Week 12
  Imaging of the head and neck will be performed using positron emission magnetic resonance imaging. MRI of the salivary glands in Sjogren's syndrome patient demonstrate inhomogeneity of the parenchyma on both T1- and T2-weighted sequences.
Change in FDG uptake on PET/MRI imaging | Baseline and Week 12
  Imaging of the head and neck will be performed using positron emission magnetic resonance imaging. FDG-PET may demonstrate areas of uptake signaling active inflammation.
Change in EULAR Sjögren's syndrome (SS) disease activity index | Baseline and Week 12
  The ESSDAI is a systemic disease activity index that was designed to measure disease activity in patients with primary Sjogren's syndrome.
  The ESSDAI consists of a composite numerical score of 12 organ specific "domains" contributing to disease activity (constitutional, lymphadenopathy, glandular, articular, cutaneous, pulmonary, renal, peripheral nervous system, central nervous system, muscular, hematological, and biological parameters). Each domain is divided into 3 to 4 levels according to the degree of activity and scored as 0 (no activity), 1 (low activity), 2 (moderate activity), or 3 (high activity). These scores are then multiplied by an assigned weight factor, ranging from 1 to 6, with the total score ranging from 0 to 123 points. A higher score denotes more disease activity.
Change in Schirmer I test | Baseline and Week 12
  Schirmer's test is used to determine whether the eye produces enough tears to keep it moist.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Baker, MD, MS, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No